CLINICAL TRIAL: NCT02104518
Title: Evaluation of a Point-of-care G6PD Diagnostic Test
Brief Title: Evaluation of Different G6PD Testing Platforms
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Eijkman Institute for Molecular Biology (Other)
Responsible Party: Sponsor
Other Study IDs: Eijkman-69
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Glucose-6-Phosphate Dehydrogenase Deficiency
Keywords: glucose-6-phosphate dehydrogenase; point-of-care diagnostic testing
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Left-over venous blood will be spun down and buffy coat and extracted DNA will be stored in labeled tubes for later G6PD genotyping and characterization.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- G6PD testing: Blood samples will be tested for G6PD activity levels

SUMMARY:
In this study the investigators propose to evaluate the performance of several G6PD testing platforms.

DETAILED DESCRIPTION:
In this study we propose to evaluate the performance of several G6PD testing platforms. We will also determine the concordance between point-of-care G6PD tests and the spectrophotometric gold standard. This study will also access the sensitivity and specificity between the point-of-care G6PD tests. This study will take place in Indonesia, specifically in the SW Sumba region. We will enroll 700 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least five years of age
* Patient / parental consent
* Patient willing to allow donated sample to be used in future research

Exclusion Criteria:

* Patients with severe malaria or other severe illness
* Patients who received a blood transfusion in the last three months
* Patients unwilling to allow donated blood to be used in future research

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll up to 700 volunteers from the SW Sumba region in Indonesia. The SW Sumba region is inland, and isolated from other nearby villages. The general population of SW Sumba are substance farmers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Determine concordance between point-of-care tests and spectrophotometric gold standard | Six months
  Percent agreement between the quantitative results of the G6PD tests and the spectrophotometric test.

SECONDARY OUTCOMES:
Determine sensitivity and specificity of the point-of-care G6PD tests against the spectrophotometric gold standard | Six months
  This is to determine the variance of the sensitivity and specificity of different G6PD point-of-care tests compared to the gold standard.
Measure categorical accuracy of point-of-care G6PD test against by the spectrophotometric gold standard | Six months
  Percent agreement between the qualitative G6PD test and the categorical results of the spectrophotometric gold standard
Determine concordance between point-of-care G6PD tests and the florescent spot test | Six months
  Compare sensitivity & specificity of qualitative results of the G6PD test and the categorical results of the florescent spot test.
Define the G6PD-normal and deficient profiles in the SW Sumba population. | Six months
  Determine the profile of the SW Sumba area in regards to normal and deficient population spread.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Winasti Satyagraha, PhD, Study Chair — Eijkman Institute for Molecular Biology; Kevin Baird, PhD, Study Chair — Oxford University Clinical Research Unit Indonesia
Locations (1):
- Eijkman Institute for Molecular Biology, Jakarta, Indonesia